CLINICAL TRIAL: NCT03756714
Title: Safety and Performance of the TFCC FastFix in the Wrist
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TFCCFF.PMCF.2017.12
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Suture Retention Device to Facilitate Triangular Fibrocartilage Complex (TFCC) Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess safety and performance post-market of the TFCC FastFix in the wrist.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone TFCC repair using the TFCC FastFix Device
* Patients aged 18 years and older
* Patients that are > 12 months post-operative.

Exclusion Criteria:

* Subjects who are < 12 months post-operative
* Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 12 months post-operative.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had TFCC repair using TFCC FastFix device
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Rate (%) of clinical success of six months post-operative. Clinical success is defined as wrists without signs of device failure and/or re-intervention after assessment by surgeon | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Mangin, Study Chair — Smith & Nephew, Inc.
Locations (1):
- Miami Orthopedics & Sport Medicine Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No